CLINICAL TRIAL: NCT00911105
Title: Combined Application of Lenalidomide and Desamethasone in the Palliative Therapy of Patients With Multiple Myeloma
Brief Title: Non -Interventional Study-Palliative Therapy of Multiple Myeloma With a Combination of Lenalidomide and Dexamethasone
Acronym: REVLIMID-NIS
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-0810
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Non-interventional study; Lenalidomide; Dexamethasone; Observational; Time to progression; Clinical routine; Germany; Plasmacytoma
MeSH Terms: conditions — Multiple Myeloma; Plasmacytoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with multiple myeloma: Patients with multiple myeloma receiving second line therapy or higher.

SUMMARY:
Purpose of this non-interventional study is the documentation of efficacy and safety data of multiple myeloma therapy with a combined treatment of Lenalidomide and Dexamethasone in daily routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma with at least one previous therapy.
* 18 years or older
* Signed, written informed consent

Exclusion Criteria:

* Pregnancy or nursing
* All other exclusion criteria listed in SmPC (summary of product characteristics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mutiple myeloma receiving a combination therapy with Lenalidomide and Dexamethasone.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2009-05; Primary Completion 2012-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | maximum 3 years per Patient

SECONDARY OUTCOMES:
Overall Response Rate | maximum 3 years per Patient
Time to Treatment Discontinuation (TTD) | maximum 3 years per Patient
Overall Survival (OS) | maximum 3 years per Patient
Safety Profile | maximum 3 years per Patient
Dosage of Lenalidomide and Dexamethasone | maximum 3 years per Patient
Kidney Function | maximum 3 years per Patient
Neutropenia / Infection (Concomitant Medication) | maximum 3 years per Patient
Thrombosis Prophylaxis | maximum 3 years per Patient

CONTACTS AND LOCATIONS:
Locations (20):
- Germany (20):
  - Onkologische Schwerpunktpraxis, Bad Homburg
  - Onkologische Schwerpunktpraxis, Berlin
  - Onkologisches Versorgungszentrum Friedrichshain, Berlin
  - Onkologische Praxis, Berlin
  - Onkologische Gemeinschaftspraxis, Frankfurt am Main
  - Praxis für Innere Medizin, Germering
  - MedResearch - Medizinisches Studien- und Dokumentationszentrum Leipziger Land, Groitzsch
  - Internistische Gemeinschaftspraxis, Güstrow
  - Praxis für Innere Medizin, Haematologie und Internistische Onkologie, Hamburg
  - Tumorpraxis Heidenheim, Heidenheim
  - Onkol. Gem.praxis Dr. M. Neise & Dr. A. Lollert, Krefeld
  - Onkologisches Zentrum Lebach, Lebach
  - Onkologische Gemeinschaftspraxis, Lehrte
  - Gemeinschaftspraxis Dr. Aldaoud - Dr. Schwarzer, Leipzig
  - Praxis für Haematologie und Onkologie, Mühlheim
  - Praxis fuer Innere Medizin, Neumarkt I. D. O.
  - Praxis fuer Onkologie und Haematologie, Neuss
  - Haematologisch-Onkologische Gemeinschaftspraxis, Nordhorn
  - Onkologische Praxis Oldenburg, Oldenburg
  - Onkologische Gemeinschaftspraxis, Würselen